CLINICAL TRIAL: NCT05483322
Title: An Open-Label, Expanded Access Protocol of LAM-002A (Apilimod Dimeyslate Capsules), Administered to a Single Subject With C9ORF72-Associated Frontotemporal Dementia (FTD)
Brief Title: An Open-Label, Expanded Access Protocol of LAM-002A in C9ORF72-Associated Frontotemporal Dementia (FTD)
Status: No longer available | Type: Expanded Access
Sponsor: OrphAI Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: LAM-002A-FTD-EAP
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Frontotemporal Dementia
MeSH Terms: conditions — Frontotemporal Dementia | interventions — apilimod

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: LAM-002A — 25mg capsules
  Other Names: apilimod dimesylate

SUMMARY:
This is an open-label, single subject, expanded access protocol (EAP) of the LAM-002A investigational product administered orally at 125 mg BID for 52 weeks.

DETAILED DESCRIPTION:
LAM-002A will be provided for expanded access for an individual patient under 21 CFR 312.310. It will be administered BID orally at a dose of 125 mg. Assessment of safety will include clinical observations and monitoring following administration.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of C9ORF72-associated FTD with documentation of a clinical genetic test demonstrating the presence of a pathogenic repeat expansion in C9ORF72
2. Age 18 or older
3. Capable of providing informed consent at the Screening Visit and complying with study procedures throughout the study, in the Principal Investigator's opinion.
4. In the case that the subject lacks the ability to provide informed consent. Informed consent will be sought from the subject's surrogate representative.
5. Able to safely swallow study drug capsule at screening and throughout study. May use thickened substances to assist in swallowing drug.

Exclusion Criteria:

1. Clinically significant unstable medical condition (other than FTD) that would pose a risk to the subject, according to the Principal Investigator's judgment (e.g., cardiovascular instability, systemic infection, or clinically significant laboratory abnormality or ECG changes).

   1. Gastrointestinal disease (e.g., gastric or intestinal bypass surgery, jejunostomy tube, pancreatic enzyme insufficiency, malabsorption syndrome, symptomatic inflammatory bowel disease, chronic diarrheal illness, bowel obstruction) that might interfere with drug absorption or with interpretation of gastrointestinal AEs.

      Gastrostomy tube placement is allowed prophylactically or to supplement nutrition/hydration but may not be used for study drug administration.
   2. Hepatic profile showing any of the following:

   i. Serum alanine aminotransferase (ALT) >5 × upper limit of normal (ULN). ii. Serum aspartate aminotransferase (AST) >5 × ULN. iii. Serum bilirubin >1.5 × ULN. c. Renal profile showing an estimated creatinine clearance (eClCR) <30 mL/minute (with eClCR to be calculated by the method at the laboratory performing the serum creatinine test).
2. Presence of a neurodegenerative cognitive or motor syndrome (e.g., Alzheimer's disease, Parkinson's disease) not related to the C9ORF72 repeat expansion.
3. Presence of unstable psychiatric disease or substance abuse that would impair ability of the participant to provide informed consent, in the Principal Investigator's opinion.
4. Active cancer or history of cancer, except for the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years. Active cancer includes cancers with current disease manifestations or therapy that could adversely affect subject safety and longevity, create the potential for drug-drug interactions, or compromise the interpretation of study results.
5. Prior solid organ transplantation.
6. Ongoing immunosuppressive therapy including systemic or enteric corticosteroids at screening or for the duration of the trial, at the discretion of the site investigator and medical monitor.
7. Use within 14 days prior to randomization or for the duration of the trial of a strong inhibitor or inducer of cytochrome P450 (CYP) 3A4 or expected requirement for chronic use of a strong inhibitor or inducer of CYP3A4 during study therapy (see Table 2 for a l list of drugs known to be strong inhibitors or inducers of CYP3A4), at the discretion of the Principal Investigator or Sponsor.
8. Use within 14 days prior to randomization or for the duration of the trial of drug that is a moderate-to-strong substrate of CYP2C9 (including warfarin, tolbutamide, phenytoin, glimepiride) or expected requirement for chronic use of such drugs during study therapy, at the discretion of the Principal Investigator or Sponsor.
9. Use of investigational treatments for FTD (off-label use or active participation in a clinical trial) within 5 half-lives (if known) or 30 days (whichever is longer) prior to the Screening Visit.
10. Exposure at any time to any gene therapies under investigation for the treatment of FTD (off-label use or investigational).
11. If female, breastfeeding, known to be pregnant, planning to become pregnant during the study, or of child-bearing potential and unwilling to use effective contraception for the duration of the trial and for ≥30 days after discontinuing treatment.
12. Anything that would place the subject at increased risk or preclude the subject's full compliance with or completion of the study, in the Principal Investigator's opinion.
13. If the subject is being re-screened, the disqualifying condition has not been resolved, or the mandatory wash-out duration has not occurred.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult